CLINICAL TRIAL: NCT06898814
Title: The Effects of Intravenous Iron on Mobility in Elderly Patients Following Hip Fracture Surgery: a Multicentre, Parallel Group, Randomised Controlled Trial
Brief Title: The Effects of Intravenous Iron on Mobility in Elderly Patients Following Hip Fracture Surgery
Acronym: IronHip
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Soren Overgaard (Other)
Collaborators: University Hospital Bispebjerg and Frederiksberg (Other); Copenhagen University Hospital at Herlev (Other); Odense University Hospital (Other); Musculoskeletal Statistics Unit, The Parker Institute (Unknown); Svendborg Hospital (Other)
Responsible Party: Sponsor-Investigator, Soren Overgaard, Clinical Professor, DMSc, University Hospital Bispebjerg and Frederiksberg
Organization: University Hospital Bispebjerg and Frederiksberg (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IronHip Trial; 2024-515116-42-00 (EU CTIS Number)
Record Dates: First submitted 2025-02-26; First posted 2025-03-27 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Hip Fracture; Anemia
Keywords: Hip fracture; Anemia; IV Iron; Mobility; Perioperative optimisation; Randomized Controlled Trial
MeSH Terms: conditions — Hip Fractures; Anemia | interventions — ferric derisomaltose; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participant: Blinded Primary Investigators: Blinded Coordinating Investigator: Blinded Project Manager: Blinded Database Manager: Not Blinded Obtaining baseline values (dedicated staff): Blinded Department Health Care Prof. (giving intervention): Not blinded Outcome Assessor (dedicated staff): Blinded IronHip steering committee: Blinded Sponsor: Blinded Statistician: Blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active Investigational Medicinal Product (Active Comparator)
  Interventions: Drug: Ferric Derisomaltose
- Placebo (Placebo Comparator)
  Interventions: Drug: Saline (NaCl 0,9 %) (placebo)

INTERVENTIONS:
Drug: Ferric Derisomaltose — The active intervention is a single dose of Ferric Derisomaltose, 20mg/kg body weight, diluted in 100 mL isotonic sodium chloride 0.9%
  Arms: Active Investigational Medicinal Product
Drug: Saline (NaCl 0,9 %) (placebo) — Single dose of 100 mL isotonic sodium chloride 0.9%
  Arms: Placebo

SUMMARY:
The primary aim of this clinical trial is to investigate the effects of intravenous iron on recovery in mobility compared to the pre-fracture level in patients with a hip fracture

The main questions it aims to answer are:

It is hypothesize that intravenous iron will enhance gains in mobility and hereby recovery of mobility, increase hemoglobin (Hgb), lower fatigue, have a positive effect on skeletal muscles in the weeks and months after administration.

The primary objective is to compare the effect of a single dose of ferric derisomaltose (FDI) (20 mg/kg body weight) relative to placebo on patients' recovery of functional mobility, measured as the change from baseline in the New Mobility Score.

Participants will:

- Receive either a single dose of intravenous FDI (20 mg/kg body weight) (and saline) or placebo (saline) at 1-5 days after surgery.

This trial will be conducted at three hospitals in Denmark, involving an anticipated 210 participants.

ELIGIBILITY:
Inclusion Criteria:

1. 65 years of age or older
2. Acute proximal femur fracture surgery
3. A hemoglobin measurement ≤6.5 mmol/L (10.5 g/dL) on day 1 to 5 postoperatively
4. Independent prefracture indoor walking ability, indoor NMS ≥ 2
5. Ability to speak and understand Danish
6. Able to provide informed consent on the participants own behalf

Exclusion Criteria:

1. Known allergy to intravenous iron
2. Residing permanently at a nursing home
3. Hematological conditions with a risk of iron overload e.g. haemochromatosis, hemosiderosis, or where alternative treatments are necessary e.g. haematological malignancies
4. Other contraindication to iron treatment, e.g. severe liver cirrhosis and hepatitis
5. Severe uncontrolled infection as assessed by the responsible clinician (e.g. bacteraemia or sepsis)
6. Plasma sodium levels below 125 or above 150 mmol/L on the day of inclusion
7. Renal replacement therapy
8. Severe dementia assessed by physician
9. Recent intravenous iron injection, 4 weeks prior to surgery
10. Patient declared terminally ill
11. Pathologic Fracture

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2025-06-09 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-09-14 (Estimated)

PRIMARY OUTCOMES:
New Mobility Score (NMS) | Measured as the change from baseline (reported as pre-fracture NMS) in the New Mobility Score after 4, 6 and 12 weeks
  The primary outcome is to compare the effect of a single dose of FDI (20 mg/kg body weight) relative to placebo on patients' recovery of functional mobility measured with New Mobility Score. New Mobility Score is a validated patient reported outcome measurement 0-9-point score for hip fracture patients, with 9 point equal to a fully independent indoor, outdoor and during shopping walking ability and 0 point, indicating no walking ability. Higher scores indicate a better outcome.

SECONDARY OUTCOMES:
Hemoglobin | Measured at baseline, 6 and 12 weeks after intervention.
Red blood cell transfusion requirement | Measured on postoperative day (POD) 7 and POD 30
  This will be measured by the proportion of patients who receive at least one red blood cell unit and the amounts of units per patient
Fatigue, assessed using the Verbal Rating Scale for Fatigue (F-VRS) | Measured at baseline, 4, 6 and 12 weeks after intervention.
  Fatigue will be assessed using the Verbal Rating Scale for Fatigue (F-VRS). This scale, ranging from 0 to 4, measures fatigue in hip fracture patients, where 0 indicates no fatigue and 4 represents extreme fatigue.
Quality of life with EuroQol 5-Dimension 5-Level questionnaire (EQ-5D-5L ) | Measured as a retrograde baseline the weeks prior to admission and at 6 and 12 weeks after intervention
  The EQ-5D-5L questionnaire measures health-related quality of life across five dimensions, with scores ranging from 1 (no problems) to 5 (extreme problems). Higher scores indicate worse outcomes, reflecting greater health issues.
EuroQol Visual Analogue Scale (EQ VAS 0-100) | Measured as a retrograde baseline the weeks prior to admission and at 6 and 12 weeks after intervention
  The EQ VAS 0-100 (range) is a visual analogue scale where 0 represents the worst imaginable health state and 100 represents the best. Higher scores on the EQ VAS indicate a better health outcome.
Fear of falls measured with, Short Falls Efficacy Scale International (Short-FES-I) | Measured at baseline and at 6 and 12 weeks after intervention.
  Short Falls Efficacy Scale International (Short-FES-I) measures concern about falling during various activities, with scores ranging from 7 (no concern about falling) to 28 (severe concern about falling). Higher scores indicate greater concern about falling.
30 second Sit-to-Stand-Test (STS) | Measured at baseline, 6 and 12 weeks
  Participants are encouraged to stand and fully sit as many times as possible within 30 seconds, with correct form monitored by the tester. If a participant uses their arms, they score a 0, and only correctly executed stands are counted. This test assesses a wide range of ability levels. Lower score indicates worse outcome.
Activity of daily living, asessed with Barthel Index 20 | Measured as a retrograde baseline and at 6 and 12 weeks after intervention
  Barthel 20 Index measures a patient's level of independence in daily activities, with scores ranging from 0 (complete dependence) to 20 (complete independence). Higher scores indicate a better outcome, reflecting greater independence.
Pain, assessed using the Verbal Rating Scale for pain | Measured at baseline and at 6 and 12 weeks after intervention
  Hip fracture-related pain will be assessed using the Verbal Rating Scale for Pain, which ranges from 0 to 4. A score of 0 indicates no pain, while a score of 4 represents unbearable or the worst imaginable pain
Days alive and at home up to 30 (DAH30) | Measured at 6 weeks after intervention.
  The DAH30 is determined using a combination of electronic medical records (obtaining length of stay) and direct participant inquiries at the 6 week follow up
Serious adverse event (SAE) | Will be assessed up to the 6 weeks follow up
  SAE defined following the ICH - GCP guidelines
Mortality | 90 days
  The time of death is determined using validated registry-based data, from which survival rates, as well as 30-day and 90-day mortality rates, are calculated.

OTHER OUTCOMES:
A. Cost-effectiveness analysis | 90 days post intervention
  Explorative outcome A: Cost-effectiveness analysis will be made from a societal perspective including cost of FDI, hospital bed days, readmissions, outpatient visits and costs related to lost productivity of the patients (production loss). The analysis will be done according to the guidelines for health economic evaluation. The analysis will be based on data from the electronic patient records and data on the duration of patient's sick leave and absence from work from patient surveys. The main results from the analysis will be a comparison of the mean costs per patient in the intervention and the control group, the mean change in Quality Adjusted Life Years gained in the two groups (based on EQ5D) and the incremental cost-effectives ratio.
B. Physical Activity | SENS motion activity monitor measurements will be collected 10 days after the 6-week follow-up.
  Explorative outcome B: This outcome focuses on evaluating the effect of intravenous iron on 24-hour physical activity of patients. Physical activity will be measured using the SENS motion activity monitor. Each participant will wear the monitor for 10 days starting at the 6-week follow-up, measuring their time spent lying, sitting, standing, walking, and transitioning between these states. After 10 days, the monitor will be collected, and data will be analyzed to compare the combined amount of time spent standing and walking between the two groups. This outcome will be measured on the participants enrolled at Bispebjerg Hospital.
C. Hand Grip Strength | Hand grip strength will be measured at baseline and again at the 6- and 12-week follow-ups.
  Explorative outcome C: Hand grip strength will be assessed using a dynamometer measured in kilograms with a higher score representing better hand grip strength. Measured on participants enrolled at Bispebjerg Hospital. This outcome aims to determine how intravenous iron therapy influences hand grip strength, comparing the changes between the two groups.
D. Knee Extension Strength | Knee extension strength will be measured at baseline and at 6- and 12-week follow-ups.
  Explorative outcome D: Knee extension strength will be measured using a dynamometer, measured in Nm/Kg with a higher score representing better Knee extension strength. Measured on participants enrolled at Bispebjerg Hospital. The goal is to examine the effect of intravenous iron therapy on knee extension strength between the two groups at these key points.
E. Cognition assessed using, Orientation-Memory-Concentration test (OMC) | Measured at baseline, week 6 and 12 post-intervention.
  Exploratory Outcome E: Cognition will be assessed using the Orientation-Memory-Concentration (OMC) test to examine potential differences between the groups. The OMC test range from 0-28 points, with a score of 25-27 indicating no or minimal cognitive impairment, and a score of 0-7 indicating severe impairment.
F. Ferritin Levels as a Measure of Iron Status | Measured at baseline and week 6 and 12 post intervention.
  Exploratory Outcome F: This outcome focuses on assessing the ferritin levels in both the intervention and placebo groups. Ferritin will be measured in ng/mL. The aim is to determine how intravenous iron therapy affects ferritin levels in comparison to the placebo group.
G: Transferrin Saturation as a Measure of Iron Status | Transferrin saturation will be measured at baseline, and at the 6- and 12-week follow-ups.
  Explorative outcome G: Transferrin saturation, measured as a percentage, will be assessed in both the intervention and placebo groups. This outcome will evaluate how transferrin saturation is affected by intravenous iron therapy compared with placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Tekin Jones, MD, Principal Investigator — Copenhagen University Hospital Bispebjerg, Department of Orthopaedic Surgery and Traumatology
Locations (3):
- Denmark (3):
  - Department of Orthopedic Surgery and Traumatology, Bispebjerg, Copenhagen University Hospital, Copenhagen NV
  - Department of Orthopedic Surgery and Traumatology, Herlev, Copenhagen University Hospital, Herlev
  - Department of Orthopaedic Surgery, Odense and Svendborg University Hospital, Odense C

IPD SHARING:
Plan to Share IPD: Yes
Access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), will be provided to anyone who wishes to access the data.
Supporting Information: Study Protocol, SAP
Time Frame: Immediately following publication, no end date.
Access Criteria: Any researcher, affiliated to an established institution